CLINICAL TRIAL: NCT04999332
Title: A Phase II Trial of Perioperative Chemotherapy With Leucovorin, Oxaliplatin, Docetaxel and S-1 (LOTS) For Patients With Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Perioperative Leucovorin, Oxaliplatin, Docetaxel and S-1 (LOTS) For Locally Advanced Gastric or Gastroesophageal Junction Cancer
Acronym: LOTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: TTY Biopharm (Industry); Kaohsiung Veterans General Hospital. (Other); Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University Hospital (Other)
Responsible Party: Principal Investigator, YS Shan, MD, PhD, Professor, Dean of College of Medicine, National Cheng Kung University, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOTS-GC-01
Record Dates: First submitted 2021-07-08; First posted 2021-08-10 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; Effects of Chemotherapy; Toxicity Due to Chemotherapy
Keywords: Gastric cancer; Gastroesophageal junction cancer; Locally advanced; Perioperative chemotherapy; Triplet
MeSH Terms: conditions — Stomach Neoplasms | interventions — Leucovorin; Oxaliplatin; Docetaxel; S 1 (combination); titanium silicide

STUDY DESIGN:
Intervention Model Description: Single intervention arm with trial treatment
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perioperative chemotherapy with LOTS (Experimental): LOTS as one cycle:
  Leucovorin (30 mg) twice daily per oral, day 1 to 7; Oxaliplatin (85 mg per square meter) intravenously, day 1; Docetaxel (40 mg per square meter) intravenously, day 1; S-1 (35 mg per square meter) twice daily per oral, day 1 to 7
  Pre-operative part:
  Four cycles of LOTS every two weeks
  Operative part:
  Curative gastrectomy or gastroesophagectomy plus D2 lymphadenectomy
  Post-operative part:
  Four cycles of LOTS every two weeks
  Interventions: Drug: leucovorin, oxaliplatin, docetaxel, S-1

INTERVENTIONS:
Drug: leucovorin, oxaliplatin, docetaxel, S-1 — Perioperative chemotherapy with LOTS
  Other Names: leucovorin (Folina tab, TTY Biopharm, TW); oxaliplatin (Oxalip, TTY Biopharm, TW); docetaxel (Taxotere, Sanofi-Aventis, FR); S-1 (TS-1, Taiho, JP)

SUMMARY:
The aim of the trial is to investigate the clinical efficacy and toxicity of perioperative chemotherapy with leucovorin, oxaliplatin, docetaxel and S-1 (LOTS) in patients with locally advanced gastric or gastroesophageal junction adenocarcinoma who receive a curative surgery.

DETAILED DESCRIPTION:
The study is an open-label, single-arm, single-country and multi-center phase II investigator-initiated trial. Patients with locally advanced gastric or gastroesophageal junction adenocarcinoma who enroll the trial will receive perioperative chemotherapy with LOTS (14 days as a cycle) 4 cycles every 2 weeks, followed by operation and another 4 cycles every 2 weeks post-operatively. The primary outcome is pathological response or curative resection rate. The secondary outcome includes recurrence-free survival, overall survival, disease control rate, protocol completion rate and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have histologically-confirmed gastric or gastroesophageal junction (classified as Siewert type III) adenocarcinoma with a clinical stage of T3 or above, lymph node involvement (N+) or both according to American Joint Cancer Committee staging system, 8th edition (AJCC 8th).
2. Subjects present with at least one measurable lesion which can be accurately assessed by conventional techniques at least 2.0 cm or 1.0 cm by computed tomography (CT) or magnetic resonance imaging (MRI).
3. Subjects have a lymph node-positive disease in which that at least one of the nodes with a diameter greater or equal to 0.8 cm in the long axis. If subjects do not have a node-positive disease, a clinical stage of T3 or above and a measurable tumor is required for inclusion.
4. Subjects are above 20 years of age with an Eastern Cooperative Oncology Group (ECOG) performance status ≤1, have a life expectancy >3 months, have surgically resectable disease and are physically competent and willing to receive a curative operation.
5. Subjects have adequate organ functions, including bone marrow reserve with a leukocyte count ≥3,000 /µL and platelet count ≥100,000 /µL, hepatic reserve with a serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times of upper limits and total bilirubin ≤2.0 mg/dL, renal reserve with a creatinine clearance ≥60 mL/min and cardiac reserve with a left ventricular ejection fraction (LVEF) ≥50% by echocardiography at baseline.
6. Subjects have, or agree to establish a vascular access that permits systemic intravenous chemotherapy and are capable of ingesting capsules per oral.
7. Subjects with reproductive potentials are willing to accept contraceptive measures during the trial.
8. Subjects are functionally and cognitively capable to be informed of the trial contents and objectives (including obtaining blood and tumor tissue for the trial investigation), and agree to sign the written consent for enrollment.

Exclusion Criteria:

1. Subjects have metastatic (M1, including washing cytology positive for peritoneal carcinomatosis), recurrent gastric/gastroesophageal junction cancer (defined by an interval time less than five years from the current diagnosis to the prior initial disease), or any other underlying primary malignancies excluding carcinoma in situ or resectable skin cancer.
2. Subjects have received chemotherapies within 2 years, or a major abdominal surgery or radiotherapy within 4 weeks before the trial enrollment.
3. Subjects are known to be allergic to any of the studied chemotherapeutics.
4. Subjects have underlying chronic illnesses, including cardiopulmonary diseases, ischemic heart disease, inflammatory bowel disease, poorly-controlled diabetes mellitus, liver cirrhosis and/or peripheral neuropathy of any etiologies.
5. Subjects have active bacterial, viral, fungal or mycobacterial infections that require systemic therapy, including active infection with human immunodeficiency virus (HIV), hepatitis B or C virus (HBV or HCV)
6. Subjects are planning to conceive or already in pregnancy or breastfeeding.
7. Subjects are currently participating in any other clinical trials or studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response | after pre-operative chemotherapy and curative surgery (Week 11 to 13)
  the tumor pathological response after pre-operative chemotherapy with LOTS plus curative surgery. The pathological response is defined by tumor evaluation of complete, partial or no response according to tumor regression grading (TRG)
Curative resection rate | after pre-operative chemotherapy and curative surgery (Week 11 to 13)
  the rate of margin-free (R0) resection in the absence of macro- or microscopic residual tumors remaining at the primary tumor bed

SECONDARY OUTCOMES:
Recurrence-free survival | From date of the initiation of trial treatment until the date of disease recurrence, progression or death at any causes, whichever came first, assessed up to 48 months
  the time interval from the initiation of trial treatment to disease recurrence, progression or death at any causes
Overall survival | From date of the initiation of trial treatment until the date of death at any causes, assessed up to 48 months
  the time interval from the initiation of trial treatment to death at any causes
Disease control rate | From date of the initiation of trial treatment until the date of recurrence/death events, withdrawal from the trial at any causes, termination/completion of the trial, whichever came first, assessed up to 48 months
  the rate of patients remaining in disease control (complete, partial response and stable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines version 1.1) lasting at least three months
Protocol completion rate | From date of the initiation of trial treatment until the date of recurrence/death events, withdrawal from the trial at any causes, termination/completion of the trial, whichever came first, assessed up to 48 months
  the rate of patients completing the pre-specified protocol treatment
Treatment-emergent adverse event rate | From date of the initiation of trial treatment until the date of recurrence/death events, withdrawal from the trial at any causes, termination/completion of the trial, whichever came first, assessed up to 48 months
  the rate of protocol treatment-emergent adverse events, as graded by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Chia Jui Yen, M.D., Ph.D., Study Chair — Department of Oncology, National Cheng Kung University Hospital; Yan Shen Shan, M.D., Ph.D., Study Director — Department of Surgery, National Cheng Kung University Hospital; I Shu Chen, M.D., Principal Investigator — Department of General Surgery, Kaohsiung Veterans General Hospital; Li Yuan Bai, M.D., Ph.D., Principal Investigator — Department of Hematology/Oncology, China Medical University Hospital; Ming Huang Chen, M.D., Ph.D., Principal Investigator — Department of Oncology, Taipei Veterans General Hospital
Locations (4):
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data which are processed with de-identification procedures and underlie results in a scientific publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon publication of the data to a duration of ten years
Access Criteria: Upon a formal request to the trial chairperson or chief principal investigator

REFERENCES:
- [Result] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Result] Ychou M, Boige V, Pignon JP, Conroy T, Bouche O, Lebreton G, Ducourtieux M, Bedenne L, Fabre JM, Saint-Aubert B, Geneve J, Lasser P, Rougier P. Perioperative chemotherapy compared with surgery alone for resectable gastroesophageal adenocarcinoma: an FNCLCC and FFCD multicenter phase III trial. J Clin Oncol. 2011 May 1;29(13):1715-21. doi: 10.1200/JCO.2010.33.0597. Epub 2011 Mar 28. PMID 21444866
- [Result] Al-Batran SE, Homann N, Pauligk C, Goetze TO, Meiler J, Kasper S, Kopp HG, Mayer F, Haag GM, Luley K, Lindig U, Schmiegel W, Pohl M, Stoehlmacher J, Folprecht G, Probst S, Prasnikar N, Fischbach W, Mahlberg R, Trojan J, Koenigsmann M, Martens UM, Thuss-Patience P, Egger M, Block A, Heinemann V, Illerhaus G, Moehler M, Schenk M, Kullmann F, Behringer DM, Heike M, Pink D, Teschendorf C, Lohr C, Bernhard H, Schuch G, Rethwisch V, von Weikersthal LF, Hartmann JT, Kneba M, Daum S, Schulmann K, Weniger J, Belle S, Gaiser T, Oduncu FS, Guntner M, Hozaeel W, Reichart A, Jager E, Kraus T, Monig S, Bechstein WO, Schuler M, Schmalenberg H, Hofheinz RD; FLOT4-AIO Investigators. Perioperative chemotherapy with fluorouracil plus leucovorin, oxaliplatin, and docetaxel versus fluorouracil or capecitabine plus cisplatin and epirubicin for locally advanced, resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4): a randomised, phase 2/3 trial. Lancet. 2019 May 11;393(10184):1948-1957. doi: 10.1016/S0140-6736(18)32557-1. Epub 2019 Apr 11. PMID 30982686
- [Result] Kang YK, Yook JH, Park YK, et al. LBA41 - Phase III randomized study of neoadjuvant chemotherapy (CT) with docetaxel(D), oxaliplatin(O) and S-1(S) (DOS) followed by surgery and adjuvant S-1, vs surgery and adjuvant S-1, for resectable advanced gastric cancer (GC) (PRODIGY). Annals of Oncology. 2019 2019/10/01/;30:v876-v877.
- [Result] Chiang NJ, Tsai KK, Hsiao CF, Yang SH, Hsiao HH, Shen WC, Hsu C, Lin YL, Chen JS, Shan YS, Chen LT. A multicenter, phase I/II trial of biweekly S-1, leucovorin, oxaliplatin and gemcitabine in metastatic pancreatic adenocarcinoma-TCOG T1211 study. Eur J Cancer. 2020 Jan;124:123-130. doi: 10.1016/j.ejca.2019.10.023. Epub 2019 Nov 22. PMID 31765987

DOCUMENTS (1):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04999332/Prot_000.pdf